CLINICAL TRIAL: NCT04099576
Title: Physiotherapy Combined With Therapeutic Neuroscience Education Versus Physiotherapy Alone for Patients With Chronic Low Back Pain: a Randomized Controlled Trial
Brief Title: The Effect of Therapeutic Neuroscience Education on Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Suat EREL, Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60116787-020/8825
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Chronic Low-back Pain
Keywords: therapeutic neuroscience education; chronic low back pain; kinesiophobia; pain
MeSH Terms: conditions — Kinesiophobia; Pain | interventions — Physical Therapy Modalities; Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy plus Education (Experimental): The experimental group received a three-week program consisting of 15 sessions of physiotherapy and six sessions of therapeutic neuroscience education.
  Interventions: Other: physiotherapy and education
- Control group (Active Comparator): The control group received a three-week program consisting of 15 sessions of physiotherapy alone. .
  Interventions: Other: Physiotherapy alone

INTERVENTIONS:
Other: physiotherapy and education — Hot-pack, ultrasound, trancutaneus nerve electrical stimulation (TENS) and home program exercises were applied or given to the individuals within the physiotherapy program. In addition to physiotherapy, therapeutic neuroscience education were applied to experimental group. One-to-one speech sessions focusing on pain neurophysiology were organized twice a week for three weeks. Each session lasted 40 minutes. The Therapeutic neuroscience education program included nociception, ion channel neurophysiology, central and peripheral sensitization, methods to help reduce sensitization, neuroplasticity, psychosocial factors involved in the transition from acute pain to chronic pain and behavioral, cognitive responses to pain.
  Arms: Physiotherapy plus Education
Other: Physiotherapy alone — Hot-pack, ultrasound, trancutaneus nerve electrical stimulation (TENS) and home program exercises were applied or given to the individuals within the physiotherapy program.
  Arms: Control group

SUMMARY:
Ongoing fear and catastrophization in people with chronic low back pain (CLBP) causes increased pain, disability and kinesiophobia, and decreased endurance of trunk muscles. Nowadays, recurrent low back pain complaints are increasing day by day. Besides the use of electrophysical agents and exercise in the treatment of chronic low back pain, education methods used to reduce the negative effects of psychosocial factors are important for healing.

Although there were studies about the combination of Therapeutic Neuroscience Education (TNE) with exercise in CLBP, there are no studies that combine electrophysical agents, exercise and TNE methods in the literature. Therefore, in this study, we aimed to investigate whether TNE combined with physiotherapy consisting of electrophysical modalities and home program exercise is superior to only physiotherapy in patients with CLBP.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were:

* aged between 18-60 years
* to have CLBP ˃ 3 months duration
* to have independent walking ability
* to be literate in Turkish.

Exclusion Criteria:

* to have vertebral compression fractures
* to have transitional vertebrae
* to have an underlying tumoral, rheumatologic or inflammatory disease
* to have trauma, surgical history
* to be pregnant or less than six months postpartum period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 18-60 years
Enrollment: 31 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2017-09-02 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 1 minute
  Visual Analogue Scale assessed pain severity. Visual Analog Scale is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of pain. hence the left end is usually labeled 'no pain', and the right end usually labeled 'extreme pain'. The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark by using a ruler. The scale is provided a range of scores from 0-100. High score indicates a high level of pain.
Tampa Kinesiophobia Scale | Five minutes
  Tampa Kinesiophobia Scale (TKS) evaluated kinesiophobia. TKS is a questionnaire evaluating kinesiophobia due to low back pain. The TKS questionnaire contained 17 items that assessed fear-related concepts. Each item has a four-point Likert scale with scoring options tiered from "strongly agree" to "strongly disagree" and a total score ranging from 17 to 68. Higher scores represented stronger levels of fear avoidance behavior.

SECONDARY OUTCOMES:
partial curl-up | 1 minute
  partial curl-up is an endurance test evaluating endurance of trunk flexors.
modified Sorensen tests | Five minutes
  modified Sorensen tests is an endurance test evaluating isometric endurance of trunk extansors.
Roland Morris Index | Five minutes
  Roland Morris Index (RMI) consists of 24 items related to physical functions. The questionnaire is a list of 24 statements relating to activities and the impairments of pain, appetite, mood, and sleep. A total score of the questionnaire range from 0 to 24 and a higher score indicate more severe disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University Medical Ethics Committee, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data of patients will be given in SPSS program.

REFERENCES:
- [Background] Walti P, Kool J, Luomajoki H. Short-term effect on pain and function of neurophysiological education and sensorimotor retraining compared to usual physiotherapy in patients with chronic or recurrent non-specific low back pain, a pilot randomized controlled trial. BMC Musculoskelet Disord. 2015 Apr 10;16:83. doi: 10.1186/s12891-015-0533-2. PMID 25887550